CLINICAL TRIAL: NCT06292299
Title: The PARS Study: Paediatric Advanced Respiratory Service Study - An Observational Diagnostic Feasibility Study
Acronym: PARS
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Clyde and Glasgow (Other)
Collaborators: INNOVATEUK (Unknown)
Responsible Party: Principal Investigator, Ross Langley, Dr Ross Langley, NHS Greater Clyde and Glasgow
Other Study IDs: INGN22RM471P; 10072600 (Other Grant/Funding Number: PneumoWave Ltd & Innovate UK)
Record Dates: First submitted 2024-02-26; First posted 2024-03-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sleep Disordered Breathing; Apnea of Prematurity; Respiratory Rate; Sudden Unexpected Death in Epilepsy
Keywords: Sleep Disordered Breathing; Neonatal Apnoea; Sleep Diagnostics; Wearable Device; Respiratory Rate; Respiratory Pattern; Epilepsy
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea; Sudden Unexpected Death in Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient attending for overnight cardiorespiratory polysomnography sleep study: Any patient attending the Royal Hospital for Children, Glasgow sleep laboratory for overnight cardiorespiratory polysomnography for evaluation of sleep disordered breathing. Pneumowave device will collect data from patients alongside standard clinical monitoring.
  Interventions: Device: Pneumowave
- Patients in the neonatal unit, Royal Hospital for Children, Glasgow, at risk of central apnoea: Any patient currently in the Queen Elizabeth University Hospital campus neonatal unit at risk of central apnoea receiving standard care (this may include mechanically ventilated patients). Pneumowave device will collect data from patients alongside standard clinical monitoring.
  Interventions: Device: Pneumowave
- Patients attending the epilepsy monitoirng unit for Video Telemetry: Any patient attending the Royal Hospital for Children, Glasgow Epilepsy Monitoring Unit for inpatient video-telemetry at risk of apnoea during and following seizures
  Interventions: Device: Pneumowave

INTERVENTIONS:
Device: Pneumowave — Pneumowave biosensor(s) will be be used to collect data from chest +/- abdominal movement and compared to standard clinical monitoring data

SUMMARY:
Diagnostic investigations in paediatric respiratory and sleep medicine are often challenging due to patient size (due to prematurity), tolerability, and compliance with "gold standard equipment". Children with sensory/behavioural issues, at increased risk of sleep disordered breathing (SDB), often find tolerating standard diagnostic equipment difficult. There is a need to develop non-invasive, wireless, devices designed for the paediatric population. Devices must address health in-equalities as high-risk children, with low birth weights, genetic syndromes, or complex neuro-disabilities, are often unable to undergo current investigations, particularly in sleep medicine. Prompt and accurate diagnosis of SDB is important to facilitate early intervention and improve outcomes

Infants in the neonatal period can have immature breathing control which manifests as excessive central breathing pauses, apnoea's, whilst asleep requiring oxygen therapy. There is also a risk to newborn term infants of sudden unexpected neonatal collapse, even in "low risk" babies. Diagnosis of breathing issues in babies can be challenging since babies are often too small for standard monitoring equipment. Effective monitoring and appropriate treatment of apnoea's has been shown to improve prognosis in terms of 5-year mortality and neurodevelopmental outcomes.

Children with epilepsy are at risk of epileptic apnoea during a seizure (ictal) or post-ictal apnoea following an epileptic seizure. Epileptic and post-ictal apnoea have been implicated as causes of sudden unexpected death in epilepsy (SUDEP). Epilepsy affects approx. 50 million people worldwide. The risk of SUDEP varies in different underlying causes of epilepsy but is estimated to be the cause of 1.2 deaths for every 1,000 children with epilepsy each year.

This observational study is part of a phased clinical program of research that aims to validate a small wearable biosensor developed by PneumoWave Ltd in a paediatric clinical setting with the overall primary endpoints of monitoring and assessing respiratory pattern as an aid to sleep diagnostics, and as a device to monitor apnoea in neonatal patients and children with epilepsy at risk of SUDEP.

DETAILED DESCRIPTION:
Sleep diagnostics

The investigation of sleep disordered breathing (SDB) in children can be challenging given the requirement to apply sensors/bands that measure physiological changes as part of a cardiorespiratory sleep study (CR-poly). Children with sensory/behavioural issues, who have an increased risk of SDB, often find tolerability of standard diagnostic equipment difficult. Similarly, the usefulness is limited in low weight infants. Thus, there is a need to investigate novel devices which may provide sleep diagnostic information when a CR-poly may be inappropriate or challenging. A wearable respiratory rate (RR)/effort sensor can provide continuous remote monitoring of patients and may identify abnormal breathing patterns associated with SDB.

Central apnoea and abnormal breathing patterns in neonatal patients

Babies born prematurely can often have apnoea of prematurity requiring caffeine therapy. Similarly, term (or term corrected) infants can have immature breathing control which manifests as excessive central breathing pauses whilst asleep requiring oxygen therapy. There is also a risk to newborn term infants of sudden unexpected collapse, even in "low risk" babies. Diagnosis of breathing issues in babies can be challenging since babies are often too small for standard CR-poly equipment. We aim to use the Pneumowave sensor alongside other diagnostic equipment to assess the feasibility of using this novel sensor to aid diagnosis in the post-natal period and pre-discharge from neonatal unit. Currently, newborn infants receive no standard respiratory monitoring following delivery. We aim to use the Pneumowave sensor as an indicator of altered respiratory patterns in this patient group.

Apnoeas in patients attending the epilepsy monitoring unit

Children with epilepsy are at risk of epileptic apnoea during a seizure (ictal) or post-ictal apnoea following an epileptic seizure. Epileptic and post-ictal apnoea have been implicated as causes of sudden unexpected death in epilepsy (SUDEP). Epilepsy affects approx. 50 million people worldwide. The risk of SUDEP varies in different underlying causes of epilepsy but is estimated to be the cause of 1.2 deaths for every 1,000 children with epilepsy each year. We aim to use the Pneumowave sensor alongside other diagnostic equipment to assess the feasibility of using this novel sensor to detect ictal and post-ictal apnoea in children attending inpatient EEG video-telemetry monitoring. There are no clinical or commercially-available reliable sensors to detect epileptic apnoea. We aim to use the Pneumowave sensor as an indicator of altered respiratory patterns in this patient group and assess whether data can be reliably collected in the context of an epileptic seizure.

PneumoWave Ltd Device

PneumoWave Ltd is developing a small, chest-worn, ambulatory biosensor ("Pneumowave") to detect changes in a range of respiratory metrics. This physical monitor is linked wirelessly via Bluetooth to a central monitoring systems in the form of a mobile platform app (running on a smartphone or tablet). Real-time data analysis, event detection and alert response management algorithms will eventually be are located in the hub, mobile app - they are currently in the cloud depending on the device configuration.

The proposed technology, Pneumowave device, will be used in the diagnosis, treatment and monitoring of illness, and therefore must be regulated as a Class 2 Medical Device in accordance with the regulatory framework in each country of use. To achieve this, PneumoWave Ltd first intends to develop a device capable of detecting adverse respiratory events in the hospital setting where immediate attendance to alerts is available. Further technical development will be required prior to the submission for regulatory approval of a device that is suitable for use in the community where there may be a longer time before a response is activated.

This hospital study aims to compare the PneumoWave Ltd monitoring system with the current clinical standard for such monitoring in a range of hospital-based clinical services.

The studies will observe three distinct patient groups:

Group 1: Patients attending for an overnight CR-poly Group 2: Patients who are at risk of apnoea in the neonatal unit Group 3: Patients who are at risk of apnoea in the epilpsey monitoring unti

ELIGIBILITY:
Inclusion Criteria:

Group 1 - CR-poly group

* Patient undergoing overnight CR-poly
* Age birth to >=16 years
* Are willing and able to give informed assent/consent or have available next of Kin to provide informed consent on the participant's behalf
* Able (in the Investigators opinion) to comply with all study requirements
* Can speak and read English

Group 2 - Apnoea group

* Inpatient in neonatal unit
* Age birth (from 30 weeks gestational age) to term corrected
* Parents willing and able to give informed consent
* Able (in the Investigators opinion) to comply with all study requirements
* Can speak and read English

Group 3- VT Group attending epilepsy monitoirng unit

* Inpatient receiving video-telemetry epilepsy monitoring unit
* Age birth to <16 years
* Parents willing and able to give informed consent
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Can speak and read English

Exclusion Criteria:

Group 1 - CR-poly group

* Unable to provide consent and no next of kin to provide consent on participants behalf
* Treating clinician deems patient inappropriate to be included in study

Group 2 - Apnoea group

* No next of kin to provide consent on participants behalf
* Treating clinician deems patient inappropriate to be included in study

Group 3- VT Group attending epilepsy monitoirng unit

* Unable to provide consent and no next of kin to provide consent on participants behalf
* Treating clinician deems patient inappropriate to be included in study

Ages: 1 Minute to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target number of participants in this study is 225. 75 patients who fit group 1 characteristics, 75 patients who fit group 2 characteristics and 75 patients who fit group 3 characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of collecting respiratory waveform data using Pneumowave device in patients who have (1) attended the sleep laboratory for CR- polysomnography and (2) are inpatient in neonatal unit | 2 years
  1) Length of time device in situ on patient 2) Number of times device removed by patient / other 3) Ability of device to collect data while in situ

SECONDARY OUTCOMES:
Collate respiratory data in patients who have attended the sleep laboratory for CR- poly or inpatient in neonatal unit. Respiratory data will observe: (1) Normal respiratory effort (2) Response to treatments | 2 years
  (1) Observation of waveform data from Pneumowave device and compare to: normal care vital signs and continuous monitoring vital signs extracted from patient monitors. (2) Compare Pneumowave respiratory wave patterns to clinical events: normal respiratory patterns and clinical deterioration
Collate waveform and motion artefact data in patients who have attended overnight CR-polysomnography | 2 years
  Compare respiratory waveform patterns and motion artefact data to: banded sleep diagnostic information
Collate waveform and motion artefact data in neonatal patients at risk of central apnoea | 2 years
  (1) Observation of waveform data from Pneumowave device and compare to: normal care vital signs, continuous monitoring vital signs extracted from patient monitors (2) Compare Pneumowave respiratory wave patterns to clinical events: normal respiratory patterns, clinical deterioration ,Interventions in neonatal unit
Assess the useability of Pneumowave in the opinion of the clinician, nurse and patient | 2 years
  Interview of the stakeholders on the useability of the device: Clinician, Nurse, Patient (if able to)

CONTACTS AND LOCATIONS:
Overall Officials: Ross J Langley, MBChB BSc PhD MRCPCH, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (2):
- United Kingdom (2):
  - Royal Hospital for Children, Glasgow, Glasgow, Glasgow City
  - Royal Hospital for Children, Glasgow, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other collaborators on the grant. No identifiable data will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD will be available by December 2025
Access Criteria: PneumoWave will be able to access IPD, no patient identifiable information will be shared with PneumoWave. IPD from this study will be included in a final report, presented at paediatric meetings and published in peer reviewed paediatric journals.
URL: https://www.researchdata.scot/

REFERENCES:
- [Result] Ono T, Takegawa H, Ageishi T, Takashina M, Numasaki H, Matsumoto M, Teshima T. Respiratory monitoring with an acceleration sensor. Phys Med Biol. 2011 Oct 7;56(19):6279-89. doi: 10.1088/0031-9155/56/19/008. Epub 2011 Sep 6. PMID 21896964
- [Result] Williams GW 2nd, George CA, Harvey BC, Freeman JE. A Comparison of Measurements of Change in Respiratory Status in Spontaneously Breathing Volunteers by the ExSpiron Noninvasive Respiratory Volume Monitor Versus the Capnostream Capnometer. Anesth Analg. 2017 Jan;124(1):120-126. doi: 10.1213/ANE.0000000000001395. PMID 27384980
- [Result] Voscopoulos C, Brayanov J, Ladd D, Lalli M, Panasyuk A, Freeman J. Special article: evaluation of a novel noninvasive respiration monitor providing continuous measurement of minute ventilation in ambulatory subjects in a variety of clinical scenarios. Anesth Analg. 2013 Jul;117(1):91-100. doi: 10.1213/ANE.0b013e3182918098. Epub 2013 Jun 3. PMID 23733842
- [Result] Massaroni C, Nicolo A, Lo Presti D, Sacchetti M, Silvestri S, Schena E. Contact-Based Methods for Measuring Respiratory Rate. Sensors (Basel). 2019 Feb 21;19(4):908. doi: 10.3390/s19040908. PMID 30795595
- [Result] Folke M, Cernerud L, Ekstrom M, Hok B. Critical review of non-invasive respiratory monitoring in medical care. Med Biol Eng Comput. 2003 Jul;41(4):377-83. doi: 10.1007/BF02348078. PMID 12892358
- [Result] Chu M, Nguyen T, Pandey V, Zhou Y, Pham HN, Bar-Yoseph R, Radom-Aizik S, Jain R, Cooper DM, Khine M. Respiration rate and volume measurements using wearable strain sensors. NPJ Digit Med. 2019 Feb 13;2:8. doi: 10.1038/s41746-019-0083-3. eCollection 2019. PMID 31304358
- [Derived] Vennard H, Buchan E, Miller J, Kelly S, Cowan C, Meredith O, Henderson B, Lowe DJ, Patel N, Zuberi S, Langley R. Respiratory monitoring and apnoea detection in paediatric and neonatal patients using a wearable accelerometer-based chest sensor: protocol for an observational diagnostic feasibility study. BMJ Open. 2025 Aug 31;15(8):e104363. doi: 10.1136/bmjopen-2025-104363. PMID 40887117